CLINICAL TRIAL: NCT00338000
Title: An Open-Label Study of the Optimization of Anemia Management of EPREX (Epoetin Alfa) in Predialysis Patients With Chronic Renal Failure
Brief Title: EPO-BUL-01 - Study of the Optimization of Anemia Management of EPREX (Epoetin Alfa) in Predialysis Patients With Chronic Renal Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR012034
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Last update posted 2011-02-01 (Estimated); Status verified 2011-01

CONDITIONS: Chronic Renal Failure
Keywords: Chronic renal failure; left ventricular hypertrophy; epoetin alfa
MeSH Terms: conditions — Kidney Failure, Chronic; Hypertrophy, Left Ventricular | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: Epoetin alfa

SUMMARY:
The purpose of the study is to evaluate the effectiveness, safety and clinical outcome of Epoetin alfa with dosing regime in accordance with Summary of Product Characteristics in the treatment of anemia in predialysis.

DETAILED DESCRIPTION:
Open-label, non-randomized, multicenter study for anemic patients with hemoglobin <or=11 g/dl. The dose of epoetin alfa is the routine dosage regimen and is in accordance of the approved SmPC. That's why the study had in general two phases - first period: subcutaneous administration and second period:intravenous administration. The evaluation is made in 4 visits:baseline, 2 month (Visit 1), 4 month (Visit 2), 6 month (Visit 3), 9 month (Visit 4). Echographic evaluation - on baseline visit, Visit 3 and Visit 4.Baseline visit - weight, arterial pressure, Hemoglobin, Hematocrit, Erythrocytes, Middle Cells Volume, Middle Cells Hemoglobin, Middle Cells Hemoglobin Concentration, Transferrin, Creatinine, Clerans, Visit1, Visit 2, Visit 3, Visit 4 - Hemoglobin, Hematocrit, Erythrocytes, Middle Cells Volume, Middle Cells Hemoglobin, Middle Cells Hemoglobin Concentration. The dosage is in routine dosing regimen, the starting dose of epoetin alfa is 50 Units/kg body weight. The maintaining dose depends on hematological results. Administration - subcutaneous (during the first period), intravenous (second period). Duration of the study - 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Hb<or= 11g/dl
* Females - using adequate contraceptive method

Exclusion Criteria:

* Patients with uncontrolled or severe cardiovascular disease, including recent myocardial infarction, uncontrolled hypertension or congestive heart failure
* treatment within the previous 6 months with epoetin alfa or any erythropoietin, known hypersensitivity to the product or to any of the ingredients
* patient not in line with the approved SmPC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2001-06; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Hemoglobin change - reach of target Hb levels (measured at Visit 1, 2, 3, 4)

SECONDARY OUTCOMES:
Prevention of left ventricular hypertrophy (measured at Visit 3 and 4)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V. Clinical Trial, Study Director — Janssen Pharmaceutica N.V.